CLINICAL TRIAL: NCT01289340
Title: Pain Management and Wound Healing in Partial Thickness Burn: Comparative, Post Marketing, Observational Trail Comparing Advanced Foam Dressings to Conventional Treatment.
Brief Title: Wound Healing and Pain Management in Partial Thickness Burns
Status: Withdrawn | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, dean david ed-el, MD, Rabin Medical Center
Other Study IDs: 6021rmc
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pain
Keywords: wound healing; pain; burn
MeSH Terms: conditions — Pain; Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Polymem (R): superficial burns treated with Polymem wound dressing until complete wound healing
- Biaten IBU: burns treated with Biaten IBU until complete wound healing.
- Hartmen dressing: burns treated with hartman or saline wet dressing until wound healing

SUMMARY:
the aim of the study is to compare between two advanced wound dressing and conventional dressing for the primary ER treatment of superficial partial thickness burns

ELIGIBILITY:
Inclusion Criteria:

patients with minor superficial partial thickness burns

Exclusion Criteria:

co-morbidities, pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients ages 18-40 with no co-morbidities nor pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Estimated); Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
complete wound healing | up to two to three weeks
  final burn wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Dean D Ad El, MD, Principal Investigator — Rabin medcial Center
Locations (1):
- Beilinson hospital, RMC, Petah Tikva, Israel